CLINICAL TRIAL: NCT02035397
Title: Treatment of Morbid Obesity by Intragastric Injections of Botulinum Toxin A. A Randomized, Double-blind, Placebo Controlled, Phase II-trial
Brief Title: Intragastric Injections of Botox for the Treatment of Obesity
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013/1597; 2012-004381-18 (EudraCT Number)
Record Dates: First submitted 2014-01-12; First posted 2014-01-14 (Estimated); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Obesity, Morbid
Keywords: botulinum toxin; Endoscopy; Satiation; Diet; Weight Loss
MeSH Terms: conditions — Obesity, Morbid; Weight Loss | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin A (Experimental): Botulinum toxin type A injection in muscles of stomach wall
  Interventions: Drug: Botulinum Toxin Type A
- Saline solution (Placebo Comparator): Placebo (saline solution) injection first 6 months, then active treatment
  Interventions: Drug: Botulinum Toxin Type A; Drug: Saline solution

INTERVENTIONS:
Drug: Botulinum Toxin Type A
  Other Names: Botox
Drug: Saline solution
  Other Names: NaCl
  Arms: Saline solution

SUMMARY:
One possible angle for treating obesity could be slowing down the gastric emptying time. By prolonging the gastric emptying time, the person would ideally experience increased sensation of satiety, and in the long run reduce food intake. If such a treatment provides a clinically significant weight loss, this could be an alternative for surgical procedures, avoiding the risk for perioperative complications as well as complications in the long run.

There are now several pilot studies documenting that intragastric treatment with botulinum toxin A (BTA) can be effective, although the treatment perspective is short and do not include repeated injections. However, they demonstrate that BTA-injections are safe for the patient. The treatment is administered by endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35

Exclusion Criteria:

* Known hypersensitivity to medication
* Neuro muscular disease
* Dysphagia
* Tendency for aspiration
* Ulcus
* Use of aminoglycoside antibiotics and/or spectinomycin lately
* Previous side effects of botox injections
* Previous bariatric surgery
* Previous cancer in GI-tract
* Other obesity treatment last 12 months
* Severe eating disorder
* Hypothyroidism
* Pregnancy/brest feeding
* Reduced competence to consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Body weight | Change from baseline to 6 months; 1 year; 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bård Kulseng, MD, PhD, Principal Investigator — Norwegian University of Science and Technology, Fac MH, IKOM
Locations (1):
- St. Olavs Hospital, Trondheim University Hospital, Trondheim, Norway